CLINICAL TRIAL: NCT04029129
Title: Near Highway Pollution: From Research to Action
Brief Title: Reducing Traffic Pollution Exposure Improves Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Douglas Brugge, Professor and Chair, UConn Health
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 19X-183=1; R01ES026980 (NIH)
Record Dates: First submitted 2019-07-16; First posted 2019-07-23 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Air Pollution
Keywords: Traffic-related air pollution; Air filtration; Blood pressure; Controlled exposure

STUDY DESIGN:
Intervention Model Description: Randomized cross over trial
Who Masked: Participant
Masking Description: Participants were not told the high, medium and low exposure context, however, some aspects of the sessions might have been apparent to them since filters were running during high, but not low exposure sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High exposure (Experimental): Ambient air was allowed freely into the room.
  Interventions: Other: Air filtration and building envelop modifications
- Medium exposure (Experimental): Limited air filtration was used to partially reduce levels of pollution in the room relative to outside.
  Interventions: Other: Air filtration and building envelop modifications
- Low exposure (Experimental): Doors and windows were closed and sealed and full filtration was used to maximally reduce pollution in the room.
  Interventions: Other: Air filtration and building envelop modifications

INTERVENTIONS:
Other: Air filtration and building envelop modifications — Air filters and closing and sealing of windows and doors was used to reduce infiltration of air pollution from outdoors in rooms next to major highways at rush hour.

SUMMARY:
This randomized trial assessed the effect of modifying building envelop and level of air filtration on blood pressure over two hour exposure sessions.

DETAILED DESCRIPTION:
Living close to major roadways is associated with elevated blood pressure (BP) amongst other adverse health effects. There is growing evidence that ultrafine particles (UFP, <100 nm in diameter), which are elevated near major roads and highways, contribute to such risks. We assessed the efficacy of high efficiency particulate arrestance (HEPA) filtration and building envelope adjustment at reducing exposure to and health effects of air pollution next to major highways.

We used a randomized three-period crossover trial design to assign 77 participants (aged 40-75 and without diagnosis of hypertension) to three two-hour exposure sessions. Sessions were conducted in one of two rooms immediately adjacent to highways. High, medium and low exposures were attained by varying the degree of air exchange and amount of HEPA filtration in the room. During high exposure sessions, the room was ventilated with outdoor air and no filtration was used. During low exposure sessions, leakage of outdoor air into the room was minimized and HEPA filtration was maximized. During medium exposure sessions, a moderate amount of HEPA filtration was used (less than half of that used in low sessions). Indoor particle number and black carbon (BC) concentrations (i.e., markers of traffic-related air pollution) were monitored continuously.

During each session participants sat quietly and wore noise-cancelling headphones, while their BP was monitored every ten minutes using an ambulatory BP monitor. We monitored pulse and oxygen saturation continuously.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criterion was age 40-75 years.
* There was a preference for people who were otherwise healthy, but overweight or obese.

Exclusion Criteria:

* A history of a major cardiovascular outcome (including myocardial ischemia (MI), stroke, angina)
* Other serious health problems (current asthma or COPD)
* Taking anti-hypertensive medications
* Smoking or living with a smoker
* Cognitive impairment
* Working at a job with high combustion exposure (taxi/truck driver, restaurant cook)
* High combustion exposure in the preceding 24 hours (driving on the highway, cooking in a restaurant, driving a truck)
* Not speaking English or Chinese.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Connecticut, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Using a 3-period crossover design, 77 participants were randomized to attend. Three 2-hour-long exposure sessions separated by 1-week washout periods.
  None was excluded.
Groups:
- High Exposure (First Session) Low, Medium: Ambient air was allowed freely into the room.
- Medium Exposure (First Session) High, Low Exposure: Limited air filtration was used to partially reduce levels of pollution in the room relative to outside.
  Air filtration and building envelop modifications: Air filters and closing and sealing of windows and doors was used to reduce infiltration of air pollution from outdoors in rooms next to major highways at rush hour.
- Low Exposure (First Session) Medium, High Exposure: Doors and windows were closed and sealed and full filtration was used to maximally reduce pollution in the room.
  Air filtration and building envelop modifications: Air filters and closing and sealing of windows and doors was used to reduce infiltration of air pollution from outdoors in rooms next to major highways at rush hour.
Period: First Intervention (2 Hours)
Arm/Group | High Exposure (First Session) Low, Medium | Medium Exposure (First Session) High, Low Exposure | Low Exposure (First Session) Medium, High Exposure
Started | 30 | 28 | 19
Completed | 30 | 28 | 19
Not Completed | 0 | 0 | 0
Period: Wash Out (1 Week)
Arm/Group | High Exposure (First Session) Low, Medium | Medium Exposure (First Session) High, Low Exposure | Low Exposure (First Session) Medium, High Exposure
Started | 30 | 28 | 19
Completed | 30 | 28 | 19
Not Completed | 0 | 0 | 0
Period: Third Intervention (2 Hours)
Arm/Group | High Exposure (First Session) Low, Medium | Medium Exposure (First Session) High, Low Exposure | Low Exposure (First Session) Medium, High Exposure
Started | 30 | 28 | 19
Completed | 30 | 28 | 19
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: A linear mixed model will be used to analyze the 3-exposure, 3-period crossover design. The primary outcome measure is the change in systolic blood pressure from the beginning of each exposure session. Before calculating change scores in each exposure session, each participant's systolic blood pressure measurements will be smoothed using a 3-time-period, centered moving average.
Groups:
- High Exposure (First Session), Low, Medium Exposure: Ambient air was allowed freely into the room. Participants first received a 2-hour-long High exposure session. After a washout period of 1 week, they then received a 2-hour-long Low exposure session. After a washout period of 1 week, they then received a 2-hour-long Medium exposure session. All sessions occurred on the same day of the week.
- Medium Exposure(First Session), High, Low Exposure: Limited air filtration was used to partially reduce levels of pollution in the room relative to outside.
  Air filtration and building envelop modifications: Air filters and closing and sealing of windows and doors was used to reduce infiltration of air pollution from outdoors in rooms next to major highways at rush hour.
  Participants first received a 2-hour-long Medium exposure session. After a washout period of 1 week, they then received a 2-hour-long High exposure session. After a washout period of 1 week, they then received a 2-hour-long Low exposure session. All sessions occurred on the same day of the week.
- Low Exposure (First Session), Medium, High Exposure: Doors and windows were closed and sealed and full filtration was used to maximally reduce pollution in the room.
  Air filtration and building envelop modifications: Air filters and closing and sealing of windows and doors was used to reduce infiltration of air pollution from outdoors in rooms next to major highways at rush hour.
  Participants first received a 2-hour-long Low exposure session. After a washout period of 1 week, they then received a 2-hour-long Medium exposure session. After a washout period of 1 week, they then received a 2-hour-long High exposure session. All sessions occurred on the same day of the week.
- Total: Total of all reporting groups
Arm/Group | High Exposure (First Session), Low, Medium Exposure | Medium Exposure(First Session), High, Low Exposure | Low Exposure (First Session), Medium, High Exposure | Total
Number analyzed (Participants) | 30 | 28 | 19 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (10.5) | 63.3 (9.6) | 59.7 (10.5) | 59.7 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 22 | 12 | 61
  Male | 3 | 6 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 3
  Not Hispanic or Latino | 29 | 26 | 19 | 74
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 23 | 21 | 15 | 59
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 6 | 6 | 3 | 15
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 28 | 19 | 77
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 115.9 (14.4) | 118.6 (17.6) | 120.3 (23.4) | 118.0 (17.9)

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure (SBP)
Description: Systolic blood pressure measured with ambulatory blood pressure monitors in mmHg.
Time Frame: Over 2 hour exposure period, we measured SBP after 20 minutes with the objective to assess change in SBP in a time series of measurements over that time period.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | High Exposure | Medium Exposure | Low Exposure
Number analyzed (Participants) | 77 | 77 | 77
mmHg | 122.3 (0.8) | 120.83 (0.7) | 119.9 (0.8)

2. Secondary Outcome: Diastolic Blood Pressure (DBP)
Description: The unit of measurement, mmHg for the diastolic blood pressure.
Time Frame: Over a 2 hour exposure period with the objective to assess change in DBP measured after 10 minutes in a time series of measurements over that time period.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | High Exposure | Medium Exposure | Low Exposure
Number analyzed (Participants) | 77 | 77 | 77
mmHg | 69.9 (0.5) | 70.4 (0.5) | 71.0 (0.5)

ADVERSE EVENTS:
Time Frame: 3 weeks.
Arm/Group | High Exposure | Medium Exposure | Low Exposure
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/28 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/28 | 0/19
Other Adverse Events (participants affected / at risk) | 0/30 | 0/28 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-26): https://cdn.clinicaltrials.gov/large-docs/29/NCT04029129/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-26): https://cdn.clinicaltrials.gov/large-docs/29/NCT04029129/ICF_001.pdf